CLINICAL TRIAL: NCT04569292
Title: Clinical Course of Cancer Patients Who Contracted COVID 19 Infection: An Observational Study
Brief Title: COVID-19 Infection in Cancer Pantients
Acronym: COICA
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Ospedale Andrea Tortora di Pagani (Network)
Responsible Party: Sponsor
Other Study IDs: COICA_PAG_01
Record Dates: First submitted 2020-09-16; First posted 2020-09-29 (Actual); Last update posted 2020-09-29 (Actual); Status verified 2020-09

CONDITIONS: Covid19
Keywords: COVID-19; Oncological patients; Cancer; Coronavirus infection disease
MeSH Terms: conditions — COVID-19; Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cancer patients: * confirmation of COVID-19 in the laboratory (RT-PCR techniques);
  * suspected cases of COVID-19; clinically diagnosed based on symptoms (fever> 37.5 °, decrease in oximeter saturation by at least 5%, cough, diarrhea, otitis, dysgeusia, myalgia, arthralgia, conjunctivitis and rhinorrhea) + close contact a COVID-19 subject positive;
  * asymptomatic cases; diagnosed based on positive swab results but without symptoms
  Interventions: Other: No intervention on patients

INTERVENTIONS:
Other: No intervention on patients — No intervention on patients

SUMMARY:
It's an obsevational retrospective/prospective study. Analyzing the evolution of COVID 19 infection in cancer patients can provide interesting information in the management of these patients. For this reason, the purpose of this study is to implement a registry to describe and monitor cancer patients affected by COVID 19, the factors that are associated with an unfavorable evolution, to develop a strategy for the risk assessment of these patients and recommendations. relating to their treatment.

Particular attention will be paid to patients suffering from urological tumors because the treatment followed by the patients would seem to expose them to a greater risk when they are infected with coronavirus, furthermore, from the literature it is clear that there may be a connection between sex hormones and ACE2 levels in the plasma. In fact, the estrons up-regulate the concentration of ACE2 in the circulation and this could be the reason why women would seem more protected than men once they contract the coronavirus infection

DETAILED DESCRIPTION:
Primary objectives:

* describe cancer patients with COVID-19 and their clinical course;
* identify predictors of the most severe clinical course;
* identify prognostic factors; Secondary objectives
* Monitor patients with urological tumors with particular attention;
* Dosing parameters of inflammation such as IL-6 and IFNα;
* Measure the ACE2 levels.

Patients with oncological pathology who contracted COVID 19 infection from January 1, 2020 until the WHO declaration of the end of the pandemic will be studied.

ELIGIBILITY:
Inclusion Criteria:

* confirmation of COVID-19 in the laboratory (RT-PCR techniques);
* suspected cases of COVID-19; clinically diagnosed based on symptoms (fever> 37.5 °, decrease in oximeter saturation by at least 5%, cough, diarrhea, otitis, dysgeusia, myalgia, arthralgia, conjunctivitis and rhinorrhea) + close contact a COVID-19 subject positive;
* asymptomatic cases; diagnosed based on positive swab results but without symptoms even dead patients

Exclusion Criteria:

-

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients with oncological pathology who contracted COVID 19 infection from January 1, 2020 until the WHO declaration of the end of the pandemic will be studied.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-04 (Estimated); Study Completion 2021-08 (Estimated)

PRIMARY OUTCOMES:
describe cancer patients with COVID-19 and their clinical course | Almost 1 year
  Describing cancer patients with COVID-19 and their clinical course will help us to identify predictors of the most severe clinical course and also prognostic factors

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Di Lorenzo, Principal Investigator — Oncology Unit
Locations (1):
- Oncology Unit, Hospital Andrea Tortora, Pagani, Salerno, Italy

IPD SHARING:
Plan to Share IPD: No